CLINICAL TRIAL: NCT01110915
Title: Advisa MRI™ System Clinical Investigation
Brief Title: Advisa MRI Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdvisaMRI
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Magnetic Resonance Imaging; Cardiac Pacemaker, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI group (Experimental): Subjects randomized to the MRI group will undergo a one-hour MRI scan, including 16 individual sequences in the chest and head region, at 9-12 weeks post-implant.
  Interventions: Device: Medtronic Advisa MRI Implantable Pulse Generator (IPG); Device: Medtronic CapSureFix MRI™ active fixation MRI lead
- Control group (Active Comparator): Subjects randomized to the Control group will wait for one hour without having any MRI scan at 9-12 weeks post-implant.
  Interventions: Device: Medtronic Advisa MRI Implantable Pulse Generator (IPG); Device: Medtronic CapSureFix MRI™ active fixation MRI lead

INTERVENTIONS:
Device: Medtronic Advisa MRI Implantable Pulse Generator (IPG) — Advisa MRI IPG is a dual chamber, multi-programmable IPG indicated to restore heart rates, improve cardiac output, prevent symptoms, or protect against arrhythmias related to cardiac impulse formation or conduction disorders. The IPG is indicated for use in patients who may benefit from rate-responsive pacing to support cardiac output during varying levels of activity and has been modified for use during an MRI exam.
  Other Names: Model A2DR01; Model A3DR01
Device: Medtronic CapSureFix MRI™ active fixation MRI lead — The Medtronic CapSureFix MRI™ active fixation MRI lead is a transvenous, bipolar, silicone, steroid eluting and active fixation pacing lead. It is based on the commercially available Medtronic Model 5076 lead and has been modified for use in the MRI environment. The MRI lead is used for both atrial and ventricular applications.
  Other Names: Model 5086 MRI lead

SUMMARY:
The purpose of the Advisa MRI System clinical study is to confirm safety and effectiveness in the clinical MRI (Magnetic Resonance Imaging) environment when subjects receive MRI scans up to 2W/kg Specific Absorption Rate (SAR) without positioning restrictions (MRI scans may occur anywhere on the body including the chest).

DETAILED DESCRIPTION:
The Advisa MRI IPG is a dual chamber, multi-programmable IPG. The IPG is indicated to restore heart rates, improve cardiac output, prevent symptoms, or protect against arrhythmias related to cardiac impulse formation or conduction disorders. The IPG is indicated for use in patients who may benefit from rate-responsive pacing to support cardiac output during varying levels of activity and has been modified for use during an MRI exam.

Subjects will have required follow-up visits after implant, at 2 months, 9-12 weeks, 3 months, 4 months, 6 months and every 6 months thereafter until the study ends. The MR scans will occur at the 9-12 weeks visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a Class I or II indication for implantation of a dual chamber pacemaker according to the American College of Cardiology (ACC)/American Heart Association (AHA)/Heart Rhythm Society (HRS) guidelines
* Subjects who are able to undergo a pectoral implant
* Subjects who are able and willing to undergo elective magnetic resonance (MR) scanning without sedation
* Subjects who are geographically stable and available for follow-up at the study center for the length of the study

Exclusion Criteria:

* Subjects with a mechanical tricuspid heart valve
* Subjects with a history of significant tricuspid valvular disease
* Subjects for whom a single dose of 1.0 milligram (mg) dexamethasone acetate may be contraindicated
* Subjects who require a legally authorized representative to obtain consent
* Subjects who have a previously implanted pacemaker or implantable cardioverter defibrillator (ICD) (abandoned pacemaker and/or defibrillator leads are not permitted; however subjects with complete system explants are not excluded)
* Subjects who are immediate candidates for an ICD
* Subjects who require an indicated MR scan, other than those specifically described in the study, before the 4 months follow-up
* Subjects with previously implanted active medical devices
* Subjects with a non-MRI compatible device (such as ICDs or neurostimulators) or material implant (e.g. non-MRI compatible sternal wires, neurostimulators, biostimulators, metals or alloys)
* Subjects with medical conditions that preclude the testing required by the protocol or limit study participation
* Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during this clinical study
* Pregnant women, or women of child bearing potential and who are not on a reliable form of birth control
* Subjects with exclusion criteria required by local law (e.g. age, breastfeeding)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Advisa MRI Trial Leader, Study Chair — Medtronic
Locations (37):
- United States (11):
  - Central Coast Cardiology, Salinas, California
  - Mid Florida Cardiology, Orlando, Florida
  - Iowa Heart Center, West Des Moines, Iowa
  - Mid America Heart Institute, Kansas City, Missouri
  - Raleigh Cardiology Associates, Raleigh, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Greenville Hospital System, Greenville, South Carolina
  - Cardiology Associates of East Tennesee, Knoxville, Tennessee
  - Baylor Heart & Vascular Hosptial, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (4):
  - St. George Hospital, Kogarah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Adelaide Cardiology, Adelaide, South Australia
  - Epworth, Richmond, Victoria
- Landesklinikum St. Pölten, Sankt Pölten, Austria
- Hôpital Saint-Joseph, Gilly, Belgium
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
- France (3):
  - CHRU Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Hôpiteaux de Rouen, Rouen
  - Centre Hospitalier Universitaire Saint Étienne, Saint-Etienne
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Rostock Anstalt öffentlichen Rechts und Medizinische Fakultät der Universität, Rostock
  - Universitätsklinikum Ulm, Ulm
- Semmelweis Egyetem AOK, Budapest, Hungary
- Rambam Health Care Campus, Haifa, Israel
- Italy (2):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Complesso Ospedaliero San Filippo Neri, Roma
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis - Locatie Oosterpark, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - HagaZiekenhuis - Locatie Leyweg, The Hague
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (2):
  - Royal Bournemouth Hospital, Bournemouth
  - Wythenshawe Hospital, Manchester

REFERENCES:
- [Result] Gimbel JR, Bello D, Schmitt M, Merkely B, Schwitter J, Hayes DL, Sommer T, Schloss EJ, Chang Y, Willey S, Kanal E; Advisa MRI System Study Investigators. Randomized trial of pacemaker and lead system for safe scanning at 1.5 Tesla. Heart Rhythm. 2013 May;10(5):685-91. doi: 10.1016/j.hrthm.2013.01.022. Epub 2013 Jan 17. PMID 23333721
- [Result] Schwitter J, Kanal E, Schmitt M, Anselme F, Albert T, Hayes DL, Bello D, Toth A, Chang Y, van Osch D, Sommer T; Advisa MRI System Study Investigators. Impact of the Advisa MRI pacing system on the diagnostic quality of cardiac MR images and contraction patterns of cardiac muscle during scans: Advisa MRI randomized clinical multicenter study results. Heart Rhythm. 2013 Jun;10(6):864-72. doi: 10.1016/j.hrthm.2013.02.019. Epub 2013 Feb 19. PMID 23434621

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from June 22, 2010 to October 12, 2011. A total of 269 subjects were enrolled at 35 centers.
Pre-assignment Details: A successful implant is defined as having a complete Advisa MRI system implant(Advisa MRI implable pulse generator (IPG) and two Model 5086MRI leads). Six subjects were exited prior to randomization. Of them, 3 subjects did not have an implant attempt and 3 subjects did not have a full Advisa MRI system. All other enrolled subjects were randomized.
Groups:
- MRI Group: Subjects randomized to the MRI group underwent a one-hour MRI scan, including 16 individual sequences in the chest and head region, at 9-12 weeks post-implant.
- Control Group: Subjects randomized to the Control group waited for one hour without having any MRI scan at 9-12 weeks post-implant.
Period: Overall Study
Arm/Group | MRI Group | Control Group
Started | 177 (Subjects being randomized to the MRI group.) | 86 (Subjects being randomized to the Control group.)
Completed | 167 (Subjects completing at least 4 months of follow-up.) | 84 (Subjects completing at least 4 months of follow-up.)
Not Completed | 10 | 2
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI Group | Control Group | Total
Number analyzed (Participants) | 177 | 86 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 24 | 83
  >=65 years | 118 | 62 | 180
Age Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.8) | 68.7 (10.8) | 68.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 32 | 100
  Male | 109 | 54 | 163
Region of Enrollment [Number; unit: participants]
  United States | 35 | 17 | 52
  Australia | 15 | 5 | 20
  Canada | 5 | 3 | 8
  Europe | 112 | 56 | 168
  Middle East | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging (MRI)-Related Complications
Description: For each subject in this objective, the endpoint was the occurrence of an MRI-related complication within 30 days post-MRI. An independent Adverse Event Advisory Committee (AEAC) determined whether each adverse event was a complication and whether it was MRI-related.
Time Frame: MRI scan to one-month post-MRI scan
Population: Subjects who had an MRI scan and completed their 4-month visit (or a later follow-up), or had an MRI-related complication within one month post-MRI were included in the analysis.
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 148
participants | 0
Statistical Analysis 1: Comparison: MRI Group; Null Hypothesis: MRI-related complication rate between the MRI scan and one-month post-MRI >=10%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions — A priori threshold for statistical significance was 0.025; Percentage = 0, 97.5% CI 1-sided [upper limit 2.5]

2. Primary Outcome: Atrial Pacing Capture Threshold Success
Description: Subjects' atrial pacing capture threshold was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was when a subject experienced an increase less than or equal to 0.5V (volts) between the two visits.
Time Frame: Pre-MRI/waiting period to one month post-MRI/waiting period
Population: To be included in the analysis, subjects in the MRI group must undergo an MRI scan and those in the Control group must complete the 9-12 week visit, and all the subjects must have valid pacing capture threshold measurements at pre-MRI/waiting period and the 4-month visit.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 141 | 75
participants | 141 | 75
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group -10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; Farrington-Manning test; A priori threshold for statistical significance was 0.025. Because there were no failures in either group, a p-value could not be calculated; Difference in percentages = 0

3. Primary Outcome: Ventricular Pacing Capture Threshold Success
Description: Subjects' ventricular pacing capture threshold was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was when a subject experienced an increase less than or equal to 0.5V (volts) between the two visits.
Time Frame: Pre-MRI /waiting period to 1-month post-MRI/waiting period
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 149 | 80
participants | 146 | 78
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group -10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p < 0.0001, Farrington-Manning test — A priori threshold for statistical significance was 0.025; Difference in percentages = 0.5, 95% CI 2-sided [-5.0 to 5.9]

4. Secondary Outcome: Atrial Sensed Amplitude Success
Description: Subjects' atrial sensed amplitude was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was defined as a 50% or less decrease in atrial sensed amplitude between the two visits.
Time Frame: Pre-MRI /waiting period to 1-month post-MRI/waiting period
Population: Only subjects with measured sensed amplitude values at both pre-MRI/waiting period and the 4-month visit were used in the analysis.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 138 | 73
participants | 134 | 72
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p = 0.0010, Farrington-Manning test — A priori threshold for statistical significance was 0.05; Difference in percentages = 1.5, 95% CI 1-sided [lower limit -6.1]

5. Secondary Outcome: Ventricular Sensed Amplitude Success
Description: Subjects' ventricular sensed amplitude was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was defined as a 50% or less decrease in ventricular sensed amplitude between the two visits.
Time Frame: Pre-MRI /waiting period to 1-month post-MRI/waiting period
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 140 | 75
participants | 138 | 74
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p = 0.0001, Farrington-Manning test — A priori threshold for statistical significance was 0.05; Difference in percentages = 0.1, 95% CI 1-sided [lower limit -4.6]

6. Secondary Outcome: Occurrence of Sustained Ventricular Arrhythmias and Asystole During MRI Scans.
Description: The endpoint was the occurrence of sustained ventricular arrhythmias and asystole during MRI scans and attributable to the MR scan. Sustained ventricular arrhythmias or asystole episodes that occurred during the MRI scan was considered attributable to the MR scan if so adjudicated by the AEAC.
Time Frame: During MRI scans
Population: All subjects successfully implanted with the Advisa MRI system who underwent MRI scans were included in the analysis. All MRI scans, whether done at the 9-12 week visit in the MRI group, or done at other times in either group were included in this analysis.
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 156
participants | 0
Statistical Analysis 1: Comparison: MRI Group; Null hypothesis: the proportion of subjects with sustained ventricular arrhythmias and asystole during MRI scans >= 10%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions — A priori threshold for statistical significance was 0.05; Percentage = 0, 95% CI 1-sided [upper limit 1.9]

7. Secondary Outcome: System-related Complications
Description: Subjects with a complication related to the implanted system, which consisted of the pacemaker, leads to the right chambers of the heart (atrium and ventricle), pacemaker software, and programmer. All adverse events in the time frame were recorded at the subject's center and assessed the AEAC. The AEAC determined whether each adverse event was a complication (requiring invasive intervention), and whether the event was related to the system.
Time Frame: Implant to four months post implant
Measure: Number; unit: participants
Groups:
- Implanted Subjects: Any subject who underwent a successful implant of the Advisa MRI system.
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 263
participants | 20
Statistical Analysis 1: Comparison: Implanted Subjects; Null hypothesis: the system-related complication rate between the implant procedure and the 4-months visit >= 20%; Test type: Superiority or Other; p < 0.05, Kaplan-Meier method — A priori threshold for statistical significance was 0.05; Complication rate at 4 months = 7.7, 95% CI 1-sided [upper limit 10.9]

ADVERSE EVENTS:
Time Frame: Up to 19 months.
Description: Adverse events were collected from all the subjects enrolled in this study, including 263 randomized and 6 non-randomized subjects. Because there were no adverse events in any of the 6 non-randomized subjects, they are not included in the following summary tables for adverse events.
Arm/Group | MRI Group | Control Group
Serious Adverse Events (participants affected / at risk) | 45/177 | 21/86
Other Adverse Events (participants affected / at risk) | 10/177 | 7/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=177) | Control Group (N=86)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 2 (2) | 2 (2)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 7 (8) | 5 (7)
Device pacing issue (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Undersensing (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=177) | Control Group (N=86)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 2 (2)
Device pacing issue (General disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.